CLINICAL TRIAL: NCT06728631
Title: A Study of Candonilimab Combined With All-trans Retinoic Acid for Prevention of Oral Cancer Recurrence in Patients With High-risk Oral Precancerous Lesions.
Brief Title: Candonilimab and ATRA Acid for Prevention of Oral Cancer Recurrence in Patients With OPL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Guopei Zhu, Dr., Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024HNRT01
Record Dates: First submitted 2024-12-08; First posted 2024-12-11 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Oral Cavity Cancer; Premalignant Lesion
MeSH Terms: conditions — Mouth Neoplasms | interventions — Tretinoin; Observation

STUDY DESIGN:
Intervention Model Description: The mixed control group includes patients who have previously experienced at least one instance of oral cancer and are also diagnosed with oral precancerous lesions. These patients will undergo routine follow-up or treatments other than the interventions used in this study's experimental group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention with Candonilimab and ATRA (Experimental): Candonilimab at a dose of 6mg/kg IV Q3W will be administered until a maximum treatment duration of 1 year. All-trans retinoic acid will be administered at a dose of 25mg/m² twice daily on days 1-14, with a treatment cycle of 21 days, until a maximum treatment duration of 6 months, or until the occurrence of oral cancer or other malignancies, death, intolerable toxicity, withdrawal of informed consent, or any other reasons specified in the protocol.
  Interventions: Drug: Candonilimab and ATRA
- mixed arm (Other): Routine follow-up or treatment methods other than those in the intervention group of this study
  Interventions: Other: other treatment or observation

INTERVENTIONS:
Drug: Candonilimab and ATRA — Candonilimab at a dose of 6mg/kg IV Q3W will be administered until a maximum treatment duration of 1 year. All-trans retinoic acid will be administered at a dose of 25mg/m² twice daily on days 1-14, with a treatment cycle of 21 days, until a maximum treatment duration of 6 months, or until the occurrence of oral cancer or other malignancies, death, intolerable toxicity, withdrawal of informed consent, or any other reasons specified in the protocol.
  Arms: Intervention with Candonilimab and ATRA
Other: other treatment or observation — other treatment other than Candonilimab/ATRA or observation
  Arms: mixed arm

SUMMARY:
The aim of this study is to involve high-risk patients with a history of malignant transformation in oral potentially malignant disorders. We will use a combination of Cardunil and all-trans retinoic acid for intervention. The effectiveness and safety of the combination therapy will be evaluated in the treatment of high-risk oral potentially malignant disorders, including the prevention of oral cancer recurrence and treatment of oral potentially malignant disorders. The findings of this study will provide evidence for tertiary prevention of oral cancer and the treatment of oral potentially malignant disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years old.
2. Patients with a history of oral potentially malignant disorders and still presenting any of the following potential malignant manifestations upon oral examination: (1) oral mucosal leukoplakia, (2) oral mucosal morphological changes (thickening, proliferation, etc.), (3) gingival atrophy, dark red gums, (4) oral mucosal ulcers, (5) white tongue coating changes, (6) oral mucosal erythema, blood blisters, etc.
3. History of one occurrence of invasive oral cancer/carcinoma in situ, and have undergone curative treatment.
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0-1.
5. Adequate function of important organs and bone marrow:

   1. Hematology parameters: absolute neutrophil count (ANC) ≥ 1.5×10^9/L, platelet count (PLT) ≥ 100×10^9/L, hemoglobin (HGB) ≥ 8g/dL.
   2. Liver function: total bilirubin (TBIL) ≤ 1.5×upper limit of normal (ULN), alanine aminotransferase (ALT) and/or aspartate transferase (AST) ≤ 2.5×ULN.
   3. Renal function: serum creatinine (Cr) ≤ 1.5×ULN.
6. Written informed consent and willingness to comply with the protocol procedures and visits.

Exclusion Criteria:

1. Patients who require adjuvant treatment such as radiation therapy or chemotherapy according to the assessment based on the malignant tumor treatment guidelines after the most recent oral cancer surgery (at least meeting any of the following criteria: T3-4, N2-3, DOI > 5mm, positive surgical margins/ < 5mm).
2. Patients who have undergone a major surgery or have unhealed wounds, ulcers, or fractures within 4 weeks before the first dose of study treatment.
3. Patients who received the last dose of radiotherapy or last dose of anti-tumor treatment (chemotherapy, targeted therapy, or tumor embolization, etc.) within 4 weeks before the first dose of study treatment.
4. History of exposure to any anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibodies.
5. Concurrent participation in another interventional clinical study, unless participating in an observational (non-interventional) clinical study or in the follow-up phase of an interventional study.
6. Use of any investigational drug within 4 weeks before the first dose of study treatment.
7. Use of immunosuppressive medication within 4 weeks before the first dose of study treatment, excluding intranasal, inhaled, or topical corticosteroids or systemic corticosteroids at physiologic doses (≤ 10 mg/day prednisone or equivalent dose of other corticosteroids).
8. Vaccination with live attenuated vaccines within 4 weeks before the first dose of study treatment or planned administration during the study.
9. Active, known, or suspected autoimmune diseases or medical history of such diseases within the past 2 years (excluding vitiligo, psoriasis, alopecia, or Grave's disease that do not require systemic treatment within the past 2 years, well-controlled hypothyroidism requiring thyroid hormone replacement, and type 1 diabetes mellitus requiring insulin replacement therapy).
10. Confirmed immunodeficiency disease.
11. History of allogeneic organ transplantation (excluding corneal transplantation) or allogeneic hematopoietic stem cell transplantation.
12. Known allergy to any monoclonal antibody component.
13. Uncontrolled severe diseases.
14. Coexistence of other malignancies, except for:

    1. Cured malignancy (e.g., papillary thyroid carcinoma).
    2. Non-melanoma skin cancer or malignancy resembling melanoma with no evidence of disease recurrence after adequate treatment.
    3. Carcinoma in situ with no evidence of disease recurrence after adequate treatment.
15. Pregnant or lactating patients. 5.4 Exclusion and Withdrawal Criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
oral-cancer free survival，OCFS | 2-year

SECONDARY OUTCOMES:
clinical response rate | 2-year
  clinical response rate of oral premalignant lesions
Safety Profile | 3 months
  Adverse Events of The Treatment
Quality-of-Life | 1 year
  EORTC QLQ-C30
overall survival, OS | 2-year

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No